CLINICAL TRIAL: NCT04148677
Title: The Role of Protopine Associated With Nuciferine (Protoves M1® Syrup) in Controlling Adverse Event During HIVEC® Instillations
Brief Title: Protoves M1® Syrup in Controlling Adverse Event During HIVEC® Instillations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cardarelli Hospital (Other)
Responsible Party: Principal Investigator, Francesco Chiancone, Assistant Medical Director, Principal Investigator, Cardarelli Hospital
Other Study IDs: M1-2019
Record Dates: First submitted 2019-10-25; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Bladder Cancer; LUTS; Pain
MeSH Terms: conditions — Urinary Bladder Neoplasms; Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Protoves M1® syrup: A combination of two alkaloid, Protopine and Nuciferine
  Interventions: Dietary Supplement: Protoves M1®
- No treatment: Patients will not receive a treatment

INTERVENTIONS:
Dietary Supplement: Protoves M1® — A combination of two alkaloid, Protopine and Nuciferine (Protoves-M1 ®)
  Groups: Protoves M1® syrup

SUMMARY:
100 patients with bladder cancer whose underwent Hyperthermic Intravesical Chemotherapy (HIVEC®) will be randomized in two groups (Group A: PROTOVES M1 SYRUP, Group B: NO TREATMENT). The aim of this study will be to analyse the role of two alkaloid, Protopine and Nuciferine (Protoves-M1 ®) in the prevention and the treatment of the low and mild grade adverse events related to the use of HIVEC® instillations.

DETAILED DESCRIPTION:
100 patients with bladder cancer whose underwent Hyperthermic Intravesical Chemotherapy (HIVEC®) will be randomized in two groups (Group A: PROTOVES M1 SYRUP, Group B: NO TREATMENT). The aim of this study will be to analyse the role of two alkaloid, Protopine and Nuciferine (Protoves-M1 ®) in the prevention and the treatment of the low and mild grade adverse events related to the use of HIVEC® instillations.

At the baseline data on demographic and anthropometric features (age, weight, height, BMI), lifestyle characteristics (smoke, alcohol), any comorbidities (hypertension, diabetes mellitus, etc.) will be collected. All patients will be undergone to a clinical evaluation (comprised general, genital and urologic examination). Before starting the treatment, the following measurements will be collected: prostate volume by transrectal ultrasound, PSA, uroflowmetry (Qmax, Volume Voided, Post-Void Residual), IPSS (International Prostatic Symptoms Score) questionnaire, OverActive Bladder questionnaire-short form (OABq-SF) 6 and 13, patient perception of intensity of urgency scale (PPIUS), and visual analogue scale (VAS). PSA and IPSS will be investigated only in male pts. In addition, the patient impression of improvement will be assessed. Improvement will be evaluated with the Patient Global Impression of Improvement questionnaire (PGI-I), a validated tool to estimate the improvement or the deterioration associated to the treatment.

The primary endpoint was the evaluation of the efficacy of the therapy with Protoves-M1 in controlling of the irritative symptoms, including nocturia, urinary frequency, bladder pain, urgency and urge incontinence related to the chemo-hyperthermia treatment. The secondary endpoint evaluated was the influences of the treatment on the uroflowmetric parameters.

After 1 and 6 weeks of therapy all patients will be undergone to a clinical and instrumental evaluation : Uroflow-Qmax (ml/s), Uroflow-Volume voided (ml),Uroflow-RPM (ml), IPSS total, OAB-q SF 6, OAB-q SF 13, PPIUS, PGI-I, VAS scale will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate-and high-risk NMIBC (non-muscle invasive bladder cancer) patients.
* Therapeutic program of HIVEC® (Recirculant hyperthermic IntraVEsical chemotherapy).
* Must be able to drink a syrup.

Exclusion Criteria:

* Uncontrolled underlying diseases (ASA III or IV)
* Post void residual urine ≥ 100 ml
* Bleeding tendency
* Drug abuse
* Chronic pelvic pain
* Urinary tract infection
* Neurological disease
* Bladder lithiasis
* Renal or liver failure
* Tachycardia and heart failure.
* Male patients with lower urinary tract symptoms (LUTS) and benign prostatic hyperplasia (BPH)with abnormal values of uroflowmetry
* Male patients with lower urinary tract symptoms (LUTS) that assume medical treatment for BPH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who referred to a general hospital to receive endoscopic treatment for bladder cancer (TURB) and then the endovescical chemioprofilaxis.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
IPSS total | 1 and 6 weeks
  The International Prostate Symptom Score (I-PSS) is based on the answers to some questions concerning urinary symptoms and one question concerning quality of life.
OAB-q SF 6 | 1 and 6 weeks
  The OAB-q SF 6 is a questionnaire developed to evaluate the overactive bladder symptom and health-related quality of life.
OAB-q SF 13 | 1 and 6 weeks
  The OAB-q SF 6 is a questionnaire developed to evaluate the overactive bladder symptom and health-related quality of life.
PPIUS | 1 and 6 weeks
  The PPIUS is a questionnaire developed to evaluate the patient perception of intensity of urgency
PGI-1 | 1 and 6 weeks
  PGI-I is a validated tool to estimate the improvement or the deterioration associated to the treatment.
VAS scale | 1 and 6 weeks
  Visual analogue scales (VAS) are 10-cm lines anchored at the ends by words that define the bounds of various pain dimensions.

SECONDARY OUTCOMES:
Qmax | 1 and 6 weeks
  Qmax (ml/s) is the maximum flow rate at uroflowmetry
Volume voided | 1 and 6 weeks
  Volume voided (ml) at uroflowmetry
RPM | 1 and 6 weeks
  Post-Void residual (ml) measures the amount of urine left in the bladder after urination.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Chiancone, Principal Investigator — AORN A.Cardarelli Urology Department

REFERENCES:
- [Background] Sousa A, Pineiro I, Rodriguez S, Aparici V, Monserrat V, Neira P, Carro E, Murias C, Uribarri C. Recirculant hyperthermic IntraVEsical chemotherapy (HIVEC) in intermediate-high-risk non-muscle-invasive bladder cancer. Int J Hyperthermia. 2016 Jun;32(4):374-80. doi: 10.3109/02656736.2016.1142618. Epub 2016 Feb 25. PMID 26915466
- [Background] Ustunes L, Laekeman GM, Gozler B, Vlietinck AJ, Ozer A, Herman AG. In vitro study of the anticholinergic and antihistaminic activities of protopine and some derivatives. J Nat Prod. 1988 Sep-Oct;51(5):1021-2. doi: 10.1021/np50059a043. No abstract available. PMID 2904975
- [Background] Fedurco M, Gregorova J, Sebrlova K, Kantorova J, Pes O, Baur R, Sigel E, Taborska E. Modulatory Effects of Eschscholzia californica Alkaloids on Recombinant GABAA Receptors. Biochem Res Int. 2015;2015:617620. doi: 10.1155/2015/617620. Epub 2015 Oct 5. PMID 26509084
- [Background] Zhang C, Deng J, Liu D, Tuo X, Yu Y, Yang H, Wang N. Nuciferine Inhibits Proinflammatory Cytokines via the PPARs in LPS-Induced RAW264.7 Cells. Molecules. 2018 Oct 22;23(10):2723. doi: 10.3390/molecules23102723. PMID 30360404
- [Background] Wang MX, Zhao XJ, Chen TY, Liu YL, Jiao RQ, Zhang JH, Ma CH, Liu JH, Pan Y, Kong LD. Nuciferine Alleviates Renal Injury by Inhibiting Inflammatory Responses in Fructose-Fed Rats. J Agric Food Chem. 2016 Oct 26;64(42):7899-7910. doi: 10.1021/acs.jafc.6b03031. Epub 2016 Oct 18. PMID 27718563
- [Background] Dmochowski R. Antimuscarinic therapy in men with lower urinary tract symptoms: what is the evidence? Curr Urol Rep. 2006 Nov;7(6):462-7. doi: 10.1007/s11934-006-0055-4. PMID 17052442